CLINICAL TRIAL: NCT05643625
Title: The Effect of Instrumental Pilates and Myofascial Release on Flexibility, Muscle Strength, Dynamic Balance, Neural Tension and Pain Threshold
Brief Title: The Effect of Pilates and Myofascial Release on Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Kübra Torpi, physiotherapist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pilates Exercise
Record Dates: First submitted 2022-11-26; First posted 2022-12-09 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Health, Subjective
Keywords: pilates; myofascial release; flexibility; muscle strength
MeSH Terms: interventions — Myofascial Release Therapy; Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: randomized prospective clinical trial
Who Masked: Participant
Masking Description: Each healthy woman will be interviewed and evaluated alone, and it will be ensured that they do not coincide with other woman who may be included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise and myofascial release group (Experimental): In this study, pilates exercise and myofascial release technique will be applied for 8 weeks, 2 days a week. Participants will be evaluated at the beginning of the study, at the end of the first session and after 8 weeks.
  Interventions: Other: Pilates exercise and myofascial release
- Pilates Exercise (Active Comparator): In this study, pilates exercise will be applied for 8 weeks, 2 days a week. Participants will be evaluated at the beginning of the study, at the end of the first session and after 8 weeks.
  Interventions: Other: Pilates exercise and myofascial release

INTERVENTIONS:
Other: Pilates exercise and myofascial release — Pilates exercise and myofascial relaxation technique will be applied to the experimental group and pilates exercise will be applied to the control group.
  Other Names: Pilates exercise

SUMMARY:
The aim of this study is to compare the short and long term effects of pilates and myofascial relaxation technique on flexibility, muscle strength, dynamic balance, neural tension and pain threshold. To evaluate the effects of myofascial release technique on neural tension. To evaluate the effects of pilates on neural tension. To evaluate the effects of the protocol applied in combination with pilates and myofascial release technique in healthy women.

DETAILED DESCRIPTION:
Pilates is a synthesis of balance, breathing and movement systems that predict the unity of mind and body developed by Joseph Pilates. Breathing correctly and adequately allows more oxygen to go to all the tissues in our body. Pilates; It includes 6 key principles: breath, concentration, control, precision / accuracy, centering, rhythm / fluency. It activates every muscle in the body, gives balance and flexibility, and shapes the posture by improving the body. By correcting the posture, it protects the musculoskeletal system problems caused by the posture disorder and helps the body to be more flexible and increase the strength and endurance of the muscles. It provides control over all joint movements, especially the spine. It improves balance and coordination. Fascia is a single, inseparable connective tissue that wraps, supports, protects, connects all tissues. It is a dynamic structure with many sensory receptors, constantly changing and adaptable, it is the largest system in the human body. Myofascial release technique can be defined as low-intensity, long-term mechanical force applied to the myofascial complex in order to dissolve fascial adhesions, reduce pain, ensure optimal length of the muscle, and increase functionality. It has been shown that myofascial release applied to the hamstrings in healthy individuals provides an increase in the normal range of motion of the hip. The effects of Pilates and myofascial release technique on flexibility, muscle strength, dynamic balance, neural tension and pain threshold will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-50
* Be woman Having a score of 600 or more when the International Physical Activity Questionnaire (Short) was administered
* Not be in menopause
* Not having had lower extremity surgery
* No traumatic injury in the last 1 year

Exclusion Criteria:

* Women entering menopause
* International Physical Activity Questionnaire (Short) score less than 600
* Those who have had lower extremity surgery
* Those with traumatic injury in the last 1 year

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 26 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Assessment of popliteal angle test | 8 weeks
  It will be used to assess hamstring muscle shortness. The person lies on his back. While the non-tested leg and back are fixed on the ground, the tested hip is 90 degrees flexed and tries to extend the knee. The value measured with the goniometer is recorded.
Assessment of Weight beating lunge test | 8 weeks
  It will be used to assess gastrocnemius flexibility. In front of the wall, the person tries to contact the wall with his knee without the sole of his feet rising from the ground. The non-tested leg can stay in the desired position and put the knee on the ground. The foot is expected to be at the maximum distance from the wall so that the knee on the tested side does not break contact with the wall. The distance between the big toe and the wall is recorded.

SECONDARY OUTCOMES:
Assessment of Back leg chest dynamometer test | 8 weeks
  The feet should be on the dynamometer with the sole in full contact. The chain of the dynamometer is adjusted so that the hips and knees are slightly flexed. The person grabs the handles with his hands and pulls them towards himself without disturbing the foot contact. 3 repetitions are performed and the maximum value is recorded.
Assessment of dynamometer test | 8 weeks
  The muscle strength of the hamstring and gastro muscles will be evaluated with a hand dynamometer. The person is asked to reveal movement. At this time, resistance is given with a dynamometer. Maximum resistance is created for a few seconds. The test is repeated 3 times and the maximum value on the dynamometer is recorded.
Assessment of Slump test | 8 weeks
  This test will be used to assess femoral nerve tension. The person sits on the chair with the hips and knees at 90º. Flexes the trunk first and then the neck. He then extends the knee and dorsiflexes the ankle. The maximum angle at which the patient can dorsiflex the ankle is measured.
Assessment of Laseque test | 8 weeks
  It will be used to assess sciatic nerve tension. While the person is lying on his back, he is asked to raise his leg straight with the knee extended. The maximum lifted angle is noted. The test is repeated 3 times and the maximum value is recorded.
Assessment of algometer | 8 weeks
  Pressure algometers developed by Fischer can measure up to 10 kg in kg/cm². There is a metal rod with a 1 cm² rubber on the end. This rubber tip ensures that the applied force is transmitted to the deep tissues. The rate and precision of the indicator allows measurement of both deep and superficial trigger points. As with other methods that evaluate trigger points, the muscles must be relaxed in order to be able to measure accurately. The tip of the pressure algometer is touched at a 90° angle to the point of the most intense sensitivity and the pressure is increased until the patient verbally expresses his discomfort. The application is repeated 3 times and the average value is recorded. For the hamstring, measurements will be taken from the recommended trigger points on the semitendinosus, semimembranosus and biceps femoris. For the gastrocnemius muscle, the measurement will be taken from the medial third of the muscle and 2 cm from the most bulging part of the muscle.
Assessment of star excursion balance test | 8 weeks
  It will be used to assess dynamic balance. 4 strips cut in 2 meters length are adhered to form 45 degree angles between them. The person stands in the middle of the star shape. When stretching with the right foot, it moves clockwise, when stretching with the left foot, it moves counterclockwise. During the test, the hands should be on the waist and their position should not change. The person reaches as far as he can reach with his foot and touches the strip lightly with the tip of his finger and returns to the starting point. Then it is continued with the other line and 8 stretches are performed in this way. The tester then draws a line with a pencil at the last point he reaches to measure. The test is repeated 3 times and the other foot is switched. The distances reached are recorded.
Assessment of single leg stance test | 8 weeks
  It will be used to evaluate static balance. The non-dominant foot is lifted on the hips and the hands are placed on the leg at the other knee level. The time he held his position is recorded. The test is repeated 3 times, the most successful result is saved. The test is repeated in the same way with the eyes closed.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Kübra Torpi Ceylan, MSc PT, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri University, Istanbul, Uskudar, Turkey (Türkiye)

REFERENCES:
- [Background] Cruz-Ferreira A, Fernandes J, Laranjo L, Bernardo LM, Silva A. A systematic review of the effects of pilates method of exercise in healthy people. Arch Phys Med Rehabil. 2011 Dec;92(12):2071-81. doi: 10.1016/j.apmr.2011.06.018. Epub 2011 Oct 24. PMID 22030232
- [Background] Segal NA, Hein J, Basford JR. The effects of Pilates training on flexibility and body composition: an observational study. Arch Phys Med Rehabil. 2004 Dec;85(12):1977-81. doi: 10.1016/j.apmr.2004.01.036. PMID 15605336